CLINICAL TRIAL: NCT05036161
Title: ROX Index and ROX Vector to Predict Nasal High Flow / Continuous Positive Airway Pressure Failure in Neonates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erebouni Medical Center (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Principal Investigator, Pavel Mazmanyan, Professor, Erebouni Medical Center
Other Study IDs: N 6-2/2, 2020
Record Dates: First submitted 2021-08-09; First posted 2021-09-05 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Predictive Value of Tests
Keywords: nasal high flow; NHF; CPAP; ROX; neonatal; newborn; respiratory distress; treatment failure
MeSH Terms: conditions — Dyspnea | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Predicting treatment failure of Nasal High Flow in newborns: newborns with respiratory distress treated with NHF
  Interventions: Other: Nasal high flow
- Predicting treatment failure of Continuous Positive Airway Pressure in newborns: newborns with respiratory distress treated with CPAP
  Interventions: Other: Continuous Positive Airway Pressure

INTERVENTIONS:
Other: Nasal high flow — Newborns with respiratory distress treated with NHF.
  Groups: Predicting treatment failure of Nasal High Flow in newborns
Other: Continuous Positive Airway Pressure — Newborns with respiratory distress treated with CPAP.
  Groups: Predicting treatment failure of Continuous Positive Airway Pressure in newborns

SUMMARY:
Nasal continuous positive airway pressure (CPAP) and Nasal High Flow (NHF) therapy are two primary therapies for the treatment of respiratory distress in newborns. However, a considerable number of infants, who are initially treated with CPAP and NHF, will develop worsening respiratory failure and eventually require intubation for mechanical ventilation and the administration of surfactant. Infants who fail noninvasive respiratory therapy may suffer the consequences of delayed intubation, surfactant administration and other adverse outcomes. The most challenging decisions in the management of respiratory distress after birth is to decide when to move from a noninvasive respiratory support to invasive mechanical ventilation and give surfactant to decrease pulmonary damage and improve outcomes. There are no clinically adequate predictors of early CPAP failure at the time of admission to the neonatal intensive care unit. Many measurements have been investigated for their ability to predict CPAP failure in infants such as fraction of inspired oxygen (FiO2), partial pressure of oxygen (PaO2), PaO2/FiO2 and the stable micro bubble test as soon as possible after birth. Roca and colleagues first established the ROX index to predict the success of NHF therapy in adults with pneumonia. The ROX index combines three common measurements: FiO2, peripheral oxygen saturation (SpO2) and respiratory rate. Combining the ROX values with the change in the respiratory rate and FiO2 can indicate whether escalation is required. It was proposed that XY plot of the key components of ROX may show the direction of changes in vector form.

The investigators hypothesized that the ROX index and ROX vector can be used for predicting the failure of CPAP and NHF in neonates.

DETAILED DESCRIPTION:
The objective is to explore the usefulness of ROX index to predict treatment failure of NHF and CPAP therapies in neonates.

The primary outcome is treatment failure within 72 h after start of the therapy with NHF or CPAP

Treatment failure criteria is reached once an infant is receiving maximal therapy for their treatment (NHF 8 L/min) or CPAP 7 cm H2O plus at least one of:

1. Sustained increase in oxygen requirement ≥50% to maintain peripheral oxygen saturation (SpO2) 90%-94%.
2. Any infant requiring urgent intubation and the subsequent mechanical ventilation, as determined by the physician.

ELIGIBILITY:
Inclusion criteria:

* They are admitted to a NICU when <24 h old, AND
* The decision has been made by the attending clinician, to commence or continue (from stabilization at birth) non-invasive respiratory support (this does not include the provision of supplemental oxygen alone), AND
* They have not previously been intubated or received surfactant

Exclusion criteria:

* They immediately require intubation and ventilation (determined by attending clinician), OR
* They already satisfy 'treatment failure' criteria, OR
* They have a known major congenital anomaly or air leak

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: neonates with respiratory distress
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants requiring escalation of treatment | 72 hours
  Treatment failure criteria is reached once an infant is receiving maximal therapy for their treatment (NHF 8 L/min) or CPAP 7 cm H2O plus at least one of:
  1. Sustained increase in oxygen requirement above ≥50% to maintain peripheral oxygen saturation (SpO2) 90%-94%.
  2. Any infant requiring urgent intubation and the subsequent mechanical ventilation, as determined by the physician.

SECONDARY OUTCOMES:
Number of participants with death | Monitored for the entire stay in hospital, until discharge, up to 6 months
  Death before discharge from the hospital
Number of participants with pneumothorax | Monitored for the entire stay in hospital, until discharge, up to 6 months
  Pneumothorax determined by chest radiograph
Number of participants with Necrotizing enterocolitis stage II-III | Monitored for the entire stay in hospital, until discharge, up to 6 months
  Necrotizing enterocolitis determined by abdominal radiograph
Number of participants with Intra-ventricular hemorrhage | Monitored for the entire stay in hospital, until discharge, up to 6 months
  Intra ventricular hemorrhage confirmed by head ultrasound
Number of participants with Bronchopulmonary dysplasia | through study completion, up to 6 months
  Bronchopulmonary dysplasia
Number of participants with Cystic Periventricular Leukomalacia | Monitored for the entire stay in hospital, until discharge, up to 6 months
  Cystic Periventricular Leukomalacia confirmed by ultrasound
Number of participants with PDA needed surgical treatment | Monitored for the entire stay in hospital, until discharge, up to 6 months
  Patent ductus arteriosus
Number of participants with ROP needing laser treatment | Monitored for the entire stay in hospital, until discharge, up to 6 months
  Retinopathy of prematurity needing laser treatment
Number of participants requiring blood transfusion | Monitored for the entire stay in hospital, until discharge, up to 6 months
  Blood transfusion
total number of days on O2 / noninvasive ventilation | Monitored for the entire stay in hospital, until discharge, up to 6 months
  total number of days on O2 / noninvasive ventilation
Total number days in the hospital | Monitored for the entire stay in hospital, until discharge, up to 6 months
  Total number days in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Mazmanyan, Prof, Principal Investigator — Head of Department of Neonatology YSMU
Locations (3):
- Armenia (3):
  - Erebouni Medical Centre, NICU, Yerevan
  - Republican Institute of Reproductive Health, NICU, Yerevan
  - Research Center of Maternal and Child Health Protection NICU, Yerevan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fuchs H, Lindner W, Leiprecht A, Mendler MR, Hummler HD. Predictors of early nasal CPAP failure and effects of various intubation criteria on the rate of mechanical ventilation in preterm infants of <29 weeks gestational age. Arch Dis Child Fetal Neonatal Ed. 2011 Sep;96(5):F343-7. doi: 10.1136/adc.2010.205898. Epub 2011 Jan 30. PMID 21278432
- [Background] Roca O, Messika J, Caralt B, Garcia-de-Acilu M, Sztrymf B, Ricard JD, Masclans JR. Predicting success of high-flow nasal cannula in pneumonia patients with hypoxemic respiratory failure: The utility of the ROX index. J Crit Care. 2016 Oct;35:200-5. doi: 10.1016/j.jcrc.2016.05.022. Epub 2016 May 31. PMID 27481760
- [Background] Roca O, Caralt B, Messika J, Samper M, Sztrymf B, Hernandez G, Garcia-de-Acilu M, Frat JP, Masclans JR, Ricard JD. An Index Combining Respiratory Rate and Oxygenation to Predict Outcome of Nasal High-Flow Therapy. Am J Respir Crit Care Med. 2019 Jun 1;199(11):1368-1376. doi: 10.1164/rccm.201803-0589OC. PMID 30576221
- [Background] Tatkov S. Nasal High-Flow Therapy: Role of FiO2 in the ROX Index. Am J Respir Crit Care Med. 2019 Jul 1;200(1):115-116. doi: 10.1164/rccm.201902-0376LE. No abstract available. PMID 30896967
- [Background] Tatkov S. ROX vector to complement ROX index during nasal high flow therapy of hypoxemic patients. J Crit Care. 2020 Aug;58:129. doi: 10.1016/j.jcrc.2019.08.012. Epub 2019 Oct 18. No abstract available. PMID 31635954